CLINICAL TRIAL: NCT04183283
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of Oral Single-Doses of LY3526318 on Cinnamaldehyde-Induced Dermal Blood Flow in Healthy Females
Brief Title: A Study of LY3526318 in Healthy Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17482; J2D-MC-CVAB (Other: Eli Lilly and Company); 2019-003613-34 (EudraCT Number)
Record Dates: First submitted 2019-11-29; First posted 2019-12-03 (Actual); Results first posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LY3526318 (Experimental): 10 milligrams (mg), 30 mg and 100 mg LY3526318 administered orally in three of four study periods.
  Interventions: Drug: LY3526318
- Placebo (Placebo Comparator): Placebo administered orally in one of four study periods.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3526318 — Administered orally.
  Arms: LY3526318
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to learn more about how LY3526318 affects blood flow to the skin in healthy women. For each participant, the study will last up to 28 days and Part B will last up to 78 days, including screening and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy female participants as determined by medical history and physical examination

  --Female participants must be nonpregnant and not lactating, or of nonchildbearing potential (either surgically sterilized [for example (e.g.) tubal occlusion, hysterectomy, bilateral salpingectomy] or physiologically incapable of becoming pregnant, or postmenopausal with amenorrhea for at least 12 consecutive months)
* Must have a body-mass index of 18 to 30 kilograms per square meter, inclusive
* Must be willing to follow specific study procedures including

  * No drugs (except study drug, hormonal contraceptives) 7 days prior to each assessment and until discharge from Clinical Research Unit (CRU)
  * No chocolate, alcohol, or caffeine containing products 24 hours prior to initiation of each assessment and until discharge
  * A complete 4 hour fast (water is allowed) prior to cinnamaldehyde (CA) assessment
* Must have suitable skin characteristics for the dermal CA challenge procedures and measured through Laser Doppler Imaging (LDI)

Exclusion Criteria:

* Must not be currently enrolled in or discontinued within the last 30 days or 5 half-lives of the study drug (whichever is longer), from a clinical study involving an investigational product or any type of medical research judged not compatible with this study
* Must not have received treatment with biological agents (such as monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing
* Must not have a history or presence of medical illness including, but not limited to, any cardiovascular, hepatic, respiratory, hematological, endocrine, psychiatric or neurological disease, convulsions, or any clinically significant laboratory abnormality that would preclude study participation
* Must not have an abnormality in the 12-lead electrocardiogram (ECG) or confirmed Frederica's corrected QT interval greater than (>) 470 millisecond (msec)
* Must not have a history of clinically significant multiple or severe drug allergies or severe post-treatment hypersensitivity reactions
* Must avoid excessive tanning
* Must not use lotions, oils, depilatory preparations, makeup, or other topical treatments on the arms on a regular basis or have used any topical treatments within 7 days prior to start of the first study day
* Must not be a habitual and heavy consumer of coffee or caffeinated beverages (more than approximately 4 cups of tea, coffee, or cola drinks/day) or who cannot refrain from caffeinated beverages 24 hours prior to CA application
* Must not be drinking alcohol 24 hours prior to each assessment
* Must not be around second-hand smoke 24 hours prior to CA application or use nicotine-containing products. Ex-smokers should have ceased smoking at least 6 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Placebo,10 mg LY3526318,100 mg LY3526318,30 mg LY3526318: Period 1: Participant received placebo orally.
  Period 2: Participants received 10 milligrams (mg) LY3526318 orally.
  Period 3: Participants received 100 mg LY3526318 orally.
  Period 4: Participants received 30 mg LY3526318 orally.
- Sequence 2: 10 mg LY3526318,30 mg LY3526318, Placebo,100 mg LY3526318: Period 1: Participant received 10 mg LY3526318 orally.
  Period 2: Participants received 30 mg LY3526318 orally.
  Period 3: Participants received Placebo orally.
  Period 4: Participants received 100 mg LY3526318 orally.
- Sequence 3: 30 mg LY3526318,100 mg LY3526318,10 mg LY3526318, Placebo: Period 1: Participant received 30 mg LY3526318 orally.
  Period 2: Participants received 100 mg LY3526318 orally.
  Period 3: Participants received 10 mg LY3526318 orally.
  Period 4: Participants received Placebo orally.
- Sequence 4: 100 mg LY3526318, Placebo, 30 mg LY3526318,10 mg LY3526318: Period 1: Participant received 100 mg LY3526318 orally.
  Period 2: Participants received Placebo orally.
  Period 3: Participants received 30 mg LY3526318 orally.
  Period 4: Participants received 10 mg LY3526318 orally.
Period: Period 1
Arm/Group | Sequence 1: Placebo,10 mg LY3526318,100 mg LY3526318,30 mg LY3526318 | Sequence 2: 10 mg LY3526318,30 mg LY3526318, Placebo,100 mg LY3526318 | Sequence 3: 30 mg LY3526318,100 mg LY3526318,10 mg LY3526318, Placebo | Sequence 4: 100 mg LY3526318, Placebo, 30 mg LY3526318,10 mg LY3526318
Started | 4 | 4 | 4 | 4
Received at Least One Dose of Study Drug | 4 | 4 | 4 | 4
Completed | 4 | 3 | 4 | 4
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Period: Washout 1(14 Days)
Arm/Group | Sequence 1: Placebo,10 mg LY3526318,100 mg LY3526318,30 mg LY3526318 | Sequence 2: 10 mg LY3526318,30 mg LY3526318, Placebo,100 mg LY3526318 | Sequence 3: 30 mg LY3526318,100 mg LY3526318,10 mg LY3526318, Placebo | Sequence 4: 100 mg LY3526318, Placebo, 30 mg LY3526318,10 mg LY3526318
Started | 4 | 3 | 4 | 4
Completed | 4 | 3 | 4 | 3
Not Completed | 0 | 0 | 0 | 1
Not completed — Positive Drug Screen | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | Sequence 1: Placebo,10 mg LY3526318,100 mg LY3526318,30 mg LY3526318 | Sequence 2: 10 mg LY3526318,30 mg LY3526318, Placebo,100 mg LY3526318 | Sequence 3: 30 mg LY3526318,100 mg LY3526318,10 mg LY3526318, Placebo | Sequence 4: 100 mg LY3526318, Placebo, 30 mg LY3526318,10 mg LY3526318
Started | 4 | 3 | 4 | 3
Completed | 4 | 3 | 4 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Washout 2 (14 Days)
Arm/Group | Sequence 1: Placebo,10 mg LY3526318,100 mg LY3526318,30 mg LY3526318 | Sequence 2: 10 mg LY3526318,30 mg LY3526318, Placebo,100 mg LY3526318 | Sequence 3: 30 mg LY3526318,100 mg LY3526318,10 mg LY3526318, Placebo | Sequence 4: 100 mg LY3526318, Placebo, 30 mg LY3526318,10 mg LY3526318
Started | 4 | 3 | 4 | 3
Completed | 4 | 3 | 4 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1: Placebo,10 mg LY3526318,100 mg LY3526318,30 mg LY3526318 | Sequence 2: 10 mg LY3526318,30 mg LY3526318, Placebo,100 mg LY3526318 | Sequence 3: 30 mg LY3526318,100 mg LY3526318,10 mg LY3526318, Placebo | Sequence 4: 100 mg LY3526318, Placebo, 30 mg LY3526318,10 mg LY3526318
Started | 4 | 3 | 4 | 4 (One participant was only dosed in Period 1, Period 3 and Period 4.)
Completed | 4 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Washout 3 (14 Days)
Arm/Group | Sequence 1: Placebo,10 mg LY3526318,100 mg LY3526318,30 mg LY3526318 | Sequence 2: 10 mg LY3526318,30 mg LY3526318, Placebo,100 mg LY3526318 | Sequence 3: 30 mg LY3526318,100 mg LY3526318,10 mg LY3526318, Placebo | Sequence 4: 100 mg LY3526318, Placebo, 30 mg LY3526318,10 mg LY3526318
Started | 4 | 3 | 4 | 4
Completed | 4 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1: Placebo,10 mg LY3526318,100 mg LY3526318,30 mg LY3526318 | Sequence 2: 10 mg LY3526318,30 mg LY3526318, Placebo,100 mg LY3526318 | Sequence 3: 30 mg LY3526318,100 mg LY3526318,10 mg LY3526318, Placebo | Sequence 4: 100 mg LY3526318, Placebo, 30 mg LY3526318,10 mg LY3526318
Started | 4 | 3 | 4 | 4
Completed | 4 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- All Participants: Sequence 1:
  Period 1: Participant received placebo orally.
  Period 2: Participants received 10 mg LY3526318 orally.
  Period 3: Participants received 100 mg LY3526318 orally.
  Period 4: Participants received 30 mg LY3526318 orally.
  Sequence 2:
  Period 1: Participant received 10 mg LY3526318 orally.
  Period 2: Participants received 30 mg LY3526318 orally.
  Period 3: Participants received Placebo orally.
  Period 4: Participants received 100 mg LY3526318 orally.
  Sequence 3:
  Period 1: Participant received 30 mg LY3526318 orally.
  Period 2: Participants received 100 mg LY3526318 orally.
  Period 3: Participants received 10 mg LY3526318 orally.
  Period 4: Participants received Placebo orally.
  Sequence 4:
  Period 1: Participant received 100 mg LY3526318 orally.
  Period 2: Participants received Placebo orally.
  Period 3: Participants received 30 mg LY3526318 orally.
  Period 4: Participants received 10 mg LY3526318 orally.
Arm/Group | All Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 16

OUTCOME MEASURES:

1. Primary Outcome: Decrease in Cinnamaldehyde (CA)-Induced Dermal Blood Flow (DBF) Relative to Placebo Measured by Laser Doppler Imaging (LDI) at 3 Hours Post-dose (LDI)
Description: CA-induced DBF was measured by laser doppler imaging (LDI). Least Squares (LS) mean was determined by analysis of variance (ANOVA) model with treatment, period, sequence, time and treatment*time interaction as fixed factors and subject within sequence as a random factor.
Time Frame: 3 hours post LY3526318 dose (pre-CA challenge), 3.3 hours post LY3526318 dose (post-CA challenge)
Population: All participants who received LY3526318 or placebo at least once and had at least one reliable post-dose pharmacodynamic measurement.
Measure: Least Squares Mean (Standard Error); unit: Perfusion unit
Groups:
- Placebo: Participant received Placebo orally.
- 10 mg LY3526318: Participant received 10 mg LY3526318 orally.
- 30 mg LY3526318: Participant received 30 mg LY3526318 orally.
- 100 mg LY3526318: Participant received 100 mg LY3526318 orally.
Arm/Group | Placebo | 10 mg LY3526318 | 30 mg LY3526318 | 100 mg LY3526318
Number analyzed (Participants) | 14 | 16 | 15 | 15
Perfusion unit
  Ring/CA Concentration (conc): Vehicle, Type: Region of Interest (ROI) | -9.46 (6.45) | -6.96 (6.45) | -14.82 (6.45) | -7.78 (6.45)
  Ring/CA conc: Vehicle, Type: Entire Image | -14.22 (3.28) | -15.1 (3.28) | -12.34 (3.28) | -13.57 (3.28)
  Ring/CA conc: 3%, Type: Region of Interest) ROI | 811.66 (98.22) | 757.83 (98.22) | 771.15 (98.22) | 758.66 (98.22)
  Ring/CA conc: 3%, Type: Entire Image | 213.82 (37.75) | 177.17 (37.75) | 191.32 (37.75) | 179.95 (37.75)
  Ring/CA conc: 10% , Type: Region of Interest (ROI) | 1264.46 (88.61) | 1233.80 (88.61) | 1165.69 (88.61) | 1049.57 (88.61)
  Ring/CA conc: 10% , Type: Entire Image | 610.17 (65.79) | 606.28 (65.79) | 419.15 (65.79) | 357.93 (65.79)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3526318; Ring/CA conc: Vehicle, Type: ROI; Test type: Superiority; p = 0.75, ANOVA; Mean Difference (Final Values) = 2.49, 90% CI 2-sided [-10.66 to 15.65]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3526318; Ring/CA conc: Vehicle, Type: ROI; Test type: Superiority; p = 0.50, ANOVA; Mean Difference (Final Values) = -5.37, 90% CI 2-sided [-18.49 to 7.76]
Statistical Analysis 3: Comparison: Placebo vs 100 mg LY3526318; Ring/CA conc: Vehicle, Type: ROI; Test type: Superiority; p = 0.83, ANOVA; Mean Difference (Final Values) = 1.68, 90% CI 2-sided [-11.48 to 14.84]
Statistical Analysis 4: Comparison: Placebo vs 10 mg LY3526318; Ring/CA conc: Vehicle, Type: Entire Image; Test type: Superiority; p = 0.84, ANOVA; Mean Difference (Final Values) = -0.88, 90% CI 2-sided [-7.91 to 6.15]
Statistical Analysis 5: Comparison: Placebo vs 30 mg LY3526318; Ring/CA conc: Vehicle, Type: Entire Image; Test type: Superiority; p = 0.66, ANOVA; Mean Difference (Final Values) = 1.89, 90% CI 2-sided [-5.13 to 8.90]
Statistical Analysis 6: Comparison: Placebo vs 100 mg LY3526318; Ring/CA conc: Vehicle, Type: Entire Image; Test type: Superiority; p = 0.88, ANOVA; Mean Difference (Final Values) = 0.65, 90% CI 2-sided [-6.38 to 7.68]
Statistical Analysis 7: Comparison: Placebo vs 10 mg LY3526318; Ring/CA conc: 3% Type: ROI; Test type: Superiority; p = 0.54, ANOVA; Mean Difference (Final Values) = -53.83, 90% CI 2-sided [-200.70 to 93.05]
Statistical Analysis 8: Comparison: Placebo vs 30 mg LY3526318; Ring/CA conc: 3% Type: ROI; Test type: Superiority; p = 0.65, ANOVA; Mean Difference (Final Values) = -40.51, 90% CI 2-sided [-187.01 to 105.98]
Statistical Analysis 9: Comparison: Placebo vs 100 mg LY3526318; Ring/CA conc: 3% Type: ROI; Test type: Superiority; p = 0.55, ANOVA; Mean Difference (Final Values) = -52.99, 90% CI 2-sided [-199.87 to 93.88]
Statistical Analysis 10: Comparison: Placebo vs 10 mg LY3526318; Ring/CA conc: 3%, Type: Entire Image; Test type: Superiority; p = 0.18, ANOVA; Mean Difference (Final Values) = -36.65, 90% CI 2-sided [-81.85 to 8.56]
Statistical Analysis 11: Comparison: Placebo vs 30 mg LY3526318; Ring/CA conc: 3%, Type: Entire Image; Test type: Superiority; p = 0.41, ANOVA; Mean Difference (Final Values) = -22.49, 90% CI 2-sided [-67.58 to 22.59]
Statistical Analysis 12: Comparison: Placebo vs 100 mg LY3526318; Ring/CA conc: 3%, Type: Entire Image; Test type: Superiority; p = 0.22, ANOVA; Mean Difference (Final Values) = -33.86, 90% CI 2-sided [-79.06 to 11.34]
Statistical Analysis 13: Comparison: Placebo vs 10 mg LY3526318; Ring/CA conc: 10%, Type: ROI; Test type: Superiority; p = 0.74, ANOVA; Mean Difference (Final Values) = -30.66, 90% CI 2-sided [-183.08 to 121.76]
Statistical Analysis 14: Comparison: Placebo vs 30 mg LY3526318; Ring/CA conc: 10%, Type: ROI; Test type: Superiority; p = 0.28, ANOVA; Mean Difference (Final Values) = -98.77, 90% CI 2-sided [-250.79 to 53.25]
Statistical Analysis 15: Comparison: Placebo vs 100 mg LY3526318; Ring/CA conc: 10%, Type: ROI; Test type: Superiority; p = 0.02, ANOVA; Mean Difference (Final Values) = -214.89, 90% CI 2-sided [-367.31 to -62.48]
Statistical Analysis 16: Comparison: Placebo vs 10 mg LY3526318; Ring/CA conc: 10% , Type: Entire Image; Test type: Superiority; p = 0.93, ANOVA; Mean Difference (Final Values) = -3.89, 90% CI 2-sided [-81.44 to 73.66]
Statistical Analysis 17: Comparison: Placebo vs 30 mg LY3526318; Ring/CA conc: 10% , Type: Entire Image; Test type: Superiority; p < .0001, ANOVA; Mean Difference (Final Values) = -191.02, 90% CI 2-sided [-268.37 to -113.67]
Statistical Analysis 18: Comparison: Placebo vs 100 mg LY3526318; Ring/CA conc: 10%, Type: Entire Image; Test type: Superiority; p < .0001, ANOVA; Mean Difference (Final Values) = -252.24, 90% CI 2-sided [-329.79 to -174.68]

2. Secondary Outcome: Decrease in CA-induced Dermal Blood Flow (DBF) Relative to Placebo Measured by Laser Speckle Contrast Imaging (LSCI) at 3 Hours Post-dose (LSCI)
Description: CA-induced DBF was measured by LSCI. LS mean was determined by ANOVA model with treatment, period, sequence, time and treatment*time interaction as fixed factors and subject within sequence as a random factor.
Time Frame: 3 hours post LY3526318 dose (pre-CA challenge), 3.3 hours post LY3526318 dose (post-CA challenge)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Perfusion unit
Arm/Group | Placebo | 10 mg LY3526318 | 30 mg LY3526318 | 100 mg LY3526318
Number analyzed (Participants) | 14 | 16 | 15 | 15
Perfusion unit
  Ring/CA conc: Vehicle, Type: Region of Interest (ROI) | -18.60 (3.49) | -18.66 (3.49) | -19.19 (3.49) | -16.07 (3.49)
  Ring/CA conc: Vehicle, Type: Entire Image | -13.50 (3.61) | -14.79 (3.61) | -12.06 (3.61) | -11.66 (3.61)
  Ring/CA conc: 3%, Type: Region of Interest (ROI) | 217.47 (26.49) | 199.09 (26.49) | 214.50 (26.49) | 2017.36 (26.49)
  Ring/CA conc: 3%, Type: Entire Image | 61.23 (12.13) | 49.92 (12.13) | 58.04 (12.13) | 50.77 (12.13)
  Ring/CA conc: 10%, Type: Region of Interest (ROI) | 306.68 (16.98) | 313.96 (16.98) | 285.98 (16.98) | 271.90 (16.98)
  Ring/CA conc: 10%, Type: Entire Image | 165.07 (19.74) | 175.09 (19.74) | 111.44 (19.74) | 85.57 (19.74)
Statistical Analysis 1: Comparison: Placebo vs 10 mg LY3526318; Ring/CA conc: Vehicle, Type: ROI; Test type: Superiority; p = 0.99, ANOVA; Mean Difference (Final Values) = -0.06, 90% CI 2-sided [-8.28 to 8.15]
Statistical Analysis 2: Comparison: Placebo vs 30 mg LY3526318; Ring/CA conc: Vehicle, Type: ROI; Test type: Superiority; p = 0.91, ANOVA; Mean Difference (Final Values) = -0.59, 90% CI 2-sided [-8.78 to 7.60]
Statistical Analysis 3: Comparison: Placebo vs 100 mg LY3526318; Ring/CA conc: Vehicle, Type: ROI; Test type: Superiority; p = 0.61, ANOVA; Mean Difference (Final Values) = 2.53, 90% CI 2-sided [-5.69 to 10.74]
Statistical Analysis 4: Comparison: Placebo vs 10 mg LY3526318; Ring/CA conc: Vehicle, Type: Entire Image; Test type: Superiority; p = 0.80, ANOVA; Mean Difference (Final Values) = -1.29, 90% CI 2-sided [-9.58 to 7.00]
Statistical Analysis 5: Comparison: Placebo vs 30 mg LY3526318; Ring/CA conc: Vehicle, Type: Entire Image; Test type: Superiority; p = 0.77, ANOVA; Mean Difference (Final Values) = 1.45, 90% CI 2-sided [-6.83 to 9.72]
Statistical Analysis 6: Comparison: Placebo vs 100 mg LY3526318; Ring/CA conc: Vehicle, Type: Entire Image; Test type: Superiority; p = 0.71, ANOVA; Mean Difference (Final Values) = 1.85, 90% CI 2-sided [-6.45 to 10.14]
Statistical Analysis 7: Comparison: Placebo vs 10 mg LY3526318; Ring/CA conc: 3%, Type: ROI; Test type: Superiority; p = 0.38, ANOVA; Mean Difference (Final Values) = -18.38, 90% CI 2-sided [-53.27 to 16.51]
Statistical Analysis 8: Comparison: Placebo vs 30 mg LY3526318; Ring/CA conc: 3%, Type: ROI; Test type: Superiority; p = 0.89, ANOVA; Mean Difference (Final Values) = -2.97, 90% CI 2-sided [-37.76 to 31.83]
Statistical Analysis 9: Comparison: Placebo vs 100 mg LY3526318; Ring/CA conc: 3%, Type: ROI; Test type: Superiority; p = 0.63, ANOVA; Mean Difference (Final Values) = -10.12, 90% CI 2-sided [-45.00 to 24.77]
Statistical Analysis 10: Comparison: Placebo vs 10 mg LY3526318; Ring/CA conc: 3%, Type: Entire Image; Test type: Superiority; p = 0.21, ANOVA; Mean Difference (Final Values) = -11.31, 90% CI 2-sided [-26.21 to 3.58]
Statistical Analysis 11: Comparison: Placebo vs 30 mg LY3526318; Ring/CA conc: 3%, Type: Entire Image; Test type: Superiority; p = 0.72, ANOVA; Mean Difference (Final Values) = -3.19, 90% CI 2-sided [-18.04 to 11.67]
Statistical Analysis 12: Comparison: Placebo vs 100 mg LY3526318; Ring/CA conc: 3%, Type: Entire Image; Test type: Superiority; p = 0.25, ANOVA; Mean Difference (Final Values) = -10.46, 90% CI 2-sided [-25.35 to 4.44]
Statistical Analysis 13: Comparison: Placebo vs 10 mg LY3526318; Ring/CA conc: 10%, Type: ROI; Test type: Superiority; p = 0.69, ANOVA; Mean Difference (Final Values) = 7.27, 90% CI 2-sided [-22.71 to 37.25]
Statistical Analysis 14: Comparison: Placebo vs 30 mg LY3526318; Ring/CA conc: 10%, Type: ROI; Test type: Superiority; p = 0.25, ANOVA; Mean Difference (Final Values) = -20.70, 90% CI 2-sided [-50.60 to 9.2]
Statistical Analysis 15: Comparison: Placebo vs 100 mg LY3526318; Ring/CA conc: 10%, Type: ROI; Test type: Superiority; p = 0.06, ANOVA; Mean Difference (Final Values) = -34.79, 90% CI 2-sided [-64.77 to -4.81]
Statistical Analysis 16: Comparison: Placebo vs 10 mg LY3526318; Ring/CA conc: 10% Type: Entire Image; Test type: Superiority; p = 0.51, ANOVA; Mean Difference (Final Values) = 10.01, 90% CI 2-sided [-15.4 to 35.42]
Statistical Analysis 17: Comparison: Placebo vs 30 mg LY3526318; Ring/CA conc: 10% Type: Entire Image; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Final Values) = -53.63, 90% CI 2-sided [-78.98 to -28.29]
Statistical Analysis 18: Comparison: Placebo vs 100 mg LY3526318; Ring/CA conc: 10% Type: Entire Image; Test type: Superiority; p < .0001, ANOVA; Mean Difference (Final Values) = -79.50, 90% CI 2-sided [-104.91 to -54.09]

3. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3526318
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3526318
Time Frame: Predose, 3 hours and 24 hours after each LY3526318 dose (days 1 through 50)
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | 10 mg LY3526318 | 30 mg LY3526318 | 100 mg LY3526318
Number analyzed (Participants) | 16 | 15 | 15
nanogram*hour per milliliter (ng*h/mL) | NA (NA) — Measurement results were below Lower Limit of Quantification. | NA (NA) — Measurement results were below Lower Limit of Quantification. | NA (NA) — Measurement results were below Lower Limit of Quantification.

4. Secondary Outcome: PK: Maximum Observed Drug Concentration (Cmax) of LY3526318
Description: PK: Maximum Observed Drug Concentration (Cmax) of LY3526318
Time Frame: Predose, 3 hours and 24 hours after each LY3526318 dose (days 1 through 50)
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (ug/mL)
Arm/Group | 10 mg LY3526318 | 30 mg LY3526318 | 100 mg LY3526318
Number analyzed (Participants) | 16 | 15 | 15
micrograms per milliliter (ug/mL) | NA (NA) — Measurement results were below Lower Limit of Quantification. | NA (NA) — Measurement results were below Lower Limit of Quantification. | NA (NA) — Measurement results were below Lower Limit of Quantification.

5. Secondary Outcome: Plasma Concentrations of LY3526318 at 3 and 24 Hours
Description: Plasma Concentrations of LY3526318 at 3 and 24 Hours
Time Frame: 3 hours and 24 hours post dose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 10 mg LY3526318 | 30 mg LY3526318 | 100 mg LY3526318
Number analyzed (Participants) | 16 | 15 | 15
nanogram per milliliter (ng/mL)
  3 Hours | 231.4 (71.4) | 627.1 (92.2) | 3669.6 (55.3)
  24 Hours | 64.9 (70.5) | 138.0 (123.8) | 854.0 (84.4)

ADVERSE EVENTS:
Time Frame: Baseline Up To 50 Days
Description: All participants who received at least one dose of study drug.
Groups:
- Placebo: Participants received Placebo orally.
- LY3526318 10 mg: Participants received 10 mg LY3526318 orally.
- LY3526318 30 mg: Participants received 30 mg LY3526318 orally.
- LY3526318 100 mg: Participants received 100 mg LY3526318 orally.
Arm/Group | Placebo | LY3526318 10 mg | LY3526318 30 mg | LY3526318 100 mg
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 11/14 | 9/16 | 5/15 | 5/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | LY3526318 10 mg (N=16) | LY3526318 30 mg (N=15) | LY3526318 100 mg (N=15)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Pyuria (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 2 (3) | 2 (2) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1)
Diastolic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT04183283/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT04183283/SAP_001.pdf